CLINICAL TRIAL: NCT05892354
Title: Efficacy of Immunonutrients in Reducing Oral Mucositis in Patients With Locoregionally Advanced Nasopharyngeal Carcinoma: A Prospective, Multicenter, Randomized Controlled Clinical Trial
Brief Title: Effect of Immunonutrients on Oral Mucositis in Nasopharyngeal Carcinoma Patients After Chemoradiotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); Zhejiang Cancer Hospital (Other); Zhejiang Provincial People's Hospital (Other); Fujian Cancer Hospital (Other Government); Fujian Provincial Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); The First Affiliated Hospital of Nanchang University (Other); Second Affiliated Hospital of Nanchang University (Other); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Qingdao Central Hospital (Other); Huizhou Municipal Central Hospital (Other); Haikou People's Hospital (Other); The Second Affiliated Hospital of Hainan Medical University (Other); Zhejiang Provincial Tongde Hospital (Other); Guilin Medical University, China (Other); Liuzhou Workers' Hospital (Other Government); Wuzhou Red Cross Hospital (Other); Red Cross Hospital of Yulin City (Other); First People's Hospital of Yulin (Other); Hainan Cancer Hospital (Other)
Responsible Party: Principal Investigator, min kang, Professor, First Affiliated Hospital of Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FirstGuangxiMu3
Record Dates: First submitted 2023-04-24; First posted 2023-06-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Locally Advanced Nasopharyngeal Carcinoma
Keywords: Immunonutrition; Nasopharyngeal Carcinoma; Chemoradiotherapy; Oral Mucositis
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Stomatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunonutrition Group (Experimental): Induction chemotherapy (IC) + Concurrent chemoradiotherapy (CCRT) and enteral immunonutrition
  Patients receive gemcitabine (1000 mg/m² d1,8) and cisplatin (80mg/m² d1) every 3 weeks for 2-3 cycles before radiotherapy and then receive intensity modulated-radiotherapy (IMRT), concurrently with cisplatin (100mg/m² d1) every 3 weeks for 2-3 cycles.
  Patients receive enteral immunonutrition, Oral Impact®, Nestle, 250ml/ bottle, 2 bottles per day, from 5 days before radiotherapy to the end of radiotherapy.
  Interventions: Dietary Supplement: Enteral immunonutrition
- Control Group (Active Comparator): Induction chemotherapy+Concurrent chemoradiotherapy and standard enteral nutrition
  Patients receive gemcitabine (1000 mg/m² d1,8) and cisplatin (80mg/m² d1) every 3 weeks for 2-3 cycles before radiotherapy and then receive intensity modulated-radiotherapy (IMRT), concurrently with cisplatin(100mg/m² d1) every 3 weeks for 2-3 cycles.
  Patients receive isocaloric standard enteral nutrition formula (ENSURE®), 250 mL per administration, 3 times per day, from 5 days before radiotherapy to the end of radiotherapy. Preparation of the 250 mL dose involves adding 200 mL of potable water to a cup and slowly stirring in 52.7 g of ENSURE powder (approximately 6 scoops).
  Interventions: Dietary Supplement: Standard enteral nutrition

INTERVENTIONS:
Dietary Supplement: Enteral immunonutrition — Enteral immunonutrition (Oral Impact®, Nestle), 250ml/ bottle, 2 bottles per day, from 5 days before radiotherapy to the end of radiotherapy.
  Arms: Immunonutrition Group
Dietary Supplement: Standard enteral nutrition — Isocaloric standard enteral nutrition formula (ENSURE®)， 250 mL per administration, 3 times per day. Preparation of the 250 mL dose involves adding 200 mL of potable water to a cup and slowly stirring in 52.7 g of ENSURE powder (approximately 6 scoops).
  Arms: Control Group

SUMMARY:
The purpose of this study was to investigate the role of immunonutrion compared with standard nutrition in reducing oral mucositis in patients with locally advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
Oral mucositis is the most common adverse reaction in patients with nasopharyngeal carcinoma receiving chemoradiotherapy, of which 40-50% of patients are severe (grade 3-4). Oral mucositis usually results in pain, dysphagia, reduced feeding, and malnutrition. Severe malnutrition in turn increases the risk of severe oral mucositis. Persistent severe oral mucositis will lead to delay and interruption of treatment, impairing patients'quality of life and prognosis. It's reported that nutritional intervention can not only reduce the risk and severity of oral mucositis and improve the nutritional status of patients with head and neck tumors, but also improve patients' tolerance to radiotherapy, quality of life, and prognosis.

Immunonutrition refers to the addition of high content of immune nutrients on the basis of sufficient calories, which not only ensures the supply of nutrition, but also takes into account the effects of anti-inflammation, regulating immunity, improving treatment tolerance, improving prognosis and so on. It has been reported that, comparing with standard enteral nutrition, the incidence of severe oral mucositis and esophagitis in patients with head and neck tumors treated with immunonutrition was lower, suffering less weight loss, and the antitumor immune response was enhanced. The 3-year OS and PFS were significantly improved in patients with good compliance.

It remains to be seen whether or not NPC patients receiving chemoradiotherapy can be benifit from immunonutritional therapy. Therefore, we conducted a prospective, multi-center, randomized controlled clinical study in patients with nasopharyngeal carcinoma who received radiotherapy and chemotherapy without metastases, to further improve the quality of life and prognosis of patients with nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
2. Age 18-70 years old, male or non-pregnant women;
3. Pathologically confirmed non-keratinizing carcinoma of the nasopharynx (differentiated or undifferentiated,WHO type II or III);
4. Newly diagnosed stage III-IVa (8th AJCC/UICC stage) NPC patients;
5. The levels of major organ function meet the following criteria:

(1)Hematology: WBC ≥ 3.0 × 10^9/L, ANC ≥ 1.5 × 10^9/L, PLT ≥ 100 × 10^9/L, HGB ≥ 90 g/L; (2) Liver function: ALT, AST≤2.5 times the upper limit of normal (ULN), total bilirubin ≤ 1.5 × ULN; (3) Renal function: BUN and CRE ≤ 1.5 × ULN or an estimated glomerular filtration rate (eGFR) ≥ 60 ml/min (calculated using the Cockcroft-Gault equation); (4) Adequate coagulation function: defined as an international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times the ULN; (5) Normal levels of cardiac enzymes; 6. The patient has signed informed consent forms and is able to comply with the study's planned visits, treatment plans, and laboratory tests.

Exclusion Criteria:

1. History of investigational Oral Impact®/ENSURE® use within the month prior to enrollment;
2. Known allergy or intolerance to any component of investigational Oral Impact®/ENSURE® or related chemotherapy drugs;
3. Poor glycemic control in patients with diabetes;
4. Patients with autoimmune diseases;
5. Patients with active infections;
6. Patients who have received radiation therapy or other anti-tumor treatments in the past;
7. Patients with a history of other malignant tumors;
8. Presence of oral mucositis at baseline;
9. Malnutrition at baseline;
10. Patients who cannot eat the required amount of food at baseline and require parenteral or enteral nutrition;
11. Inability to eat soft solid foods at baseline;
12. History of human immunodeficiency virus (HIV) or active hepatitis B/C virus infection;
13. Participation in other intervention clinical studies within one month;
14. Subjects deemed by the investigator to have other factors that may force them to terminate the study, such as having other serious illnesses (including mental illnesses) that require concomitant treatment, significantly abnormal laboratory test results, or family or social factors that may affect subject safety or data collection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of severe oral mucositis | 7 weeks
  Incidence of grade 3-4 oral mucositis

SECONDARY OUTCOMES:
The latency period of severe oral mucositis | 7 weeks
  Total duration from the start of radiotherapy to the severe oral mucositis
The duration period of severe oral mucositis | 7 weeks
  The number of days of severe oral mucositis during the oral mucositis observation period
Assessment of immune state | 4 months
  T-lymphocyte subsets
Serum hypersensitive C-reactive protein (hsCRP) level | 4 months
  Change in high sensitivity C-reactive protein from baseline to end of radiotherapy
Serum Interleukin-6 (IL-6) level | 4 months
  Change in serum level of Interleukin-6 from baseline to end of radiotherapy
Hemoglobin level | 4 months
  Change in hemoglobin level from baseline to end of radiotherapy
Serum albumin level | 4 months
  Change in hemoglobin level from baseline to end of radiotherapy
Serum Pre-Albumin level | 4 months
  Change in hemoglobin level from baseline to end of radiotherapy
Nutritional risk | 4 months
  Change in nutritional risk determined by the by the nutrition risk screening-2002 (NRS-2002) from baseline to end of radiotherapy
Nutrition status | 4 months
  Change in nutritional status determined by the Patient-Generated Subjective Global Assessment (PG-SGA) from baseline to end of radiotherapy
Physical functional status | 4 months
  Changes in handgrip strength from baseline to end of radiotherapy
overall survival rate (OS) | at 2 years after randomisation
  compare OS between two groups
progression-free survival rate (PFS) | at 2 years after randomisation
  compare PFS between two groups
Locoregional recurrence free survival rate (LRRFS) | at 2 years after randomisation
  compare LRRFS between two groups
Distance metastasis-free survival rate (DMFS) | at 2 years after randomisation
  compare DMFS between two groups
Quality of life (QoL) assessed by EORTC QLQ-C30 questionnaire | 4 months
  EORTC QLQ-C30 is a specific quality of life assessment scale based on EORTC QLQ-C 30, with 35 items. All of the scales and single-item measures range from 0 to 100. A EORTC QLQ-C30 is a specific quality of life assessment scale, with 30 items. All of the scales and single-item measures range from 0 to 100. More global and functional scales is better. less symptom scales is better.
Quality of life (QoL) assessed by the EORTC-QLQ-H&N35 Questionnaire | 4 months
  EORTC QLQ-H&N35 is a specific quality of life assessment scale based on EORTC QLQ-C 30, with 35 items. All of the scales and single-item measures range from 0 to 100. High scores represent increased (worse) symptoms.
Number of participants with adverse events | up to 2 years after randomisation
  Analysis of acute and late adverse events (AEs) are evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Min Kang, M.D, Study Chair — Department of Radiation Oncology, The First Affiliated Hospital of Guangxi Medical University
Locations (20):
- China (20):
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Affiliated Cancer Hospital & Institute of Guangzhou Medical University, Guangzhou, Guangdong
  - Huizhou Municipal Central Hospital, Huizhou, Guangdong
  - The Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Liuzhou Workers Hospital, Liuchow, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Wuzhou Red Cross Hospital, Wuzhou, Guangxi
  - First People People's Hospital of Yulin City, Yulin, Guangxi
  - Red Cross Hospital of Yulin City, Yulin, Guangxi
  - Huizhou Municipal Central Hospital, Haikou, Hainan
  - The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Hainan Cancer Hospital, Haikou, Hainan
  - Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Qingdao Central Hospital, Qingdao, Shandong
  - Zhejiang Provincial Tongde Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Background] Moslemi D, Nokhandani AM, Otaghsaraei MT, Moghadamnia Y, Kazemi S, Moghadamnia AA. Management of chemo/radiation-induced oral mucositis in patients with head and neck cancer: A review of the current literature. Radiother Oncol. 2016 Jul;120(1):13-20. doi: 10.1016/j.radonc.2016.04.001. Epub 2016 Apr 21. PMID 27113797
- [Background] Liang L, Liu Z, Zhu H, Wang H, Wei Y, Ning X, Shi Z, Jiang L, Lin Z, Yan H, Wang R, Hu K. Efficacy and safety of thalidomide in preventing oral mucositis in patients with nasopharyngeal carcinoma undergoing concurrent chemoradiotherapy: A multicenter, open-label, randomized controlled trial. Cancer. 2022 Apr 1;128(7):1467-1474. doi: 10.1002/cncr.34074. Epub 2021 Dec 15. PMID 34910297
- [Background] Xia C, Jiang C, Li W, Wei J, Hong H, Li J, Feng L, Wei H, Xin H, Chen T. A Phase II Randomized Clinical Trial and Mechanistic Studies Using Improved Probiotics to Prevent Oral Mucositis Induced by Concurrent Radiotherapy and Chemotherapy in Nasopharyngeal Carcinoma. Front Immunol. 2021 Mar 24;12:618150. doi: 10.3389/fimmu.2021.618150. eCollection 2021. PMID 33841399
- [Background] Miyata H, Yano M, Yasuda T, Yamasaki M, Murakami K, Makino T, Nishiki K, Sugimura K, Motoori M, Shiraishi O, Mori M, Doki Y. Randomized study of the clinical effects of omega-3 fatty acid-containing enteral nutrition support during neoadjuvant chemotherapy on chemotherapy-related toxicity in patients with esophageal cancer. Nutrition. 2017 Jan;33:204-210. doi: 10.1016/j.nut.2016.07.004. Epub 2016 Jul 25. PMID 27644137
- [Background] Shu Z, Zeng Z, Yu B, Huang S, Hua Y, Jin T, Tao C, Wang L, Cao C, Xu Z, Jin Q, Jiang F, Feng X, Piao Y, Huang J, Chen J, Shen W, Chen X, Wu H, Wang X, Qiu R, Lu L, Chen Y. Nutritional Status and Its Association With Radiation-Induced Oral Mucositis in Patients With Nasopharyngeal Carcinoma During Radiotherapy: A Prospective Study. Front Oncol. 2020 Nov 6;10:594687. doi: 10.3389/fonc.2020.594687. eCollection 2020. PMID 33240818
- [Background] Kabarriti R, Bontempo A, Romano M, McGovern KP, Asaro A, Viswanathan S, Kalnicki S, Garg MK. The impact of dietary regimen compliance on outcomes for HNSCC patients treated with radiation therapy. Support Care Cancer. 2018 Sep;26(9):3307-3313. doi: 10.1007/s00520-018-4198-x. Epub 2018 Apr 18. PMID 29671062
- [Background] Zheng Z, Zhao X, Zhao Q, Zhang Y, Liu S, Liu Z, Meng L, Xin Y, Jiang X. The Effects of Early Nutritional Intervention on Oral Mucositis and Nutritional Status of Patients With Head and Neck Cancer Treated With Radiotherapy. Front Oncol. 2021 Feb 1;10:595632. doi: 10.3389/fonc.2020.595632. eCollection 2020. PMID 33598427
- [Background] Boisselier P, Kaminsky MC, Thezenas S, Gallocher O, Lavau-Denes S, Garcia-Ramirez M, Alfonsi M, Cupissol D, de Forges H, Janiszewski C, Geoffrois L, Sire C, Senesse P; Head and Neck Oncology and Radiotherapy Group (GORTEC). A double-blind phase III trial of immunomodulating nutritional formula during adjuvant chemoradiotherapy in head and neck cancer patients: IMPATOX. Am J Clin Nutr. 2020 Dec 10;112(6):1523-1531. doi: 10.1093/ajcn/nqaa227. PMID 32936874
- [Background] Talvas J, Garrait G, Goncalves-Mendes N, Rouanet J, Vergnaud-Gauduchon J, Kwiatkowski F, Bachmann P, Bouteloup C, Bienvenu J, Vasson MP. Immunonutrition stimulates immune functions and antioxidant defense capacities of leukocytes in radiochemotherapy-treated head & neck and esophageal cancer patients: A double-blind randomized clinical trial. Clin Nutr. 2015 Oct;34(5):810-7. doi: 10.1016/j.clnu.2014.12.002. Epub 2014 Dec 9. PMID 25575640
- [Background] Dechaphunkul T, Arundon T, Raungkhajon P, Jiratrachu R, Geater SL, Dechaphunkul A. Benefits of immunonutrition in patients with head and neck cancer receiving chemoradiation: A phase II randomized, double-blind study. Clin Nutr. 2022 Feb;41(2):433-440. doi: 10.1016/j.clnu.2021.12.035. Epub 2021 Dec 28. PMID 35007812